CLINICAL TRIAL: NCT04737109
Title: A Single Arm, Phase I/II Trial of Neoadjuvant Androgen Deprivation, Darolutamide, and Ipatasertib in Men With Localized, High Risk Prostate Cancer Big Ten Cancer Research Consortium BTCRC-GU19-404
Brief Title: Neoadjuvant Androgen Deprivation, Darolutamide, and Ipatasertib in Men With Localized, High Risk Prostate Cancer
Acronym: ADDItion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder Decision
Sponsor: David VanderWeele (Other)
Responsible Party: Sponsor-Investigator, David VanderWeele, Associate Professor, Medicine - Hematology/Oncology, Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GU19-404
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Castrate Resistant Prostate Cancer
Keywords: prostate cancer; high risk; neoadjuvant; PTEN loss; darolutamide; ipatasertib
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ipatasertib; darolutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I De-Escalation Cohort: ADT + Ipatasertib + Darolutamide (Experimental): Cycle 0 Days 1-7: Ipatasertib Monotherapy + Androgen Deprivation Therapy (ADT) Cycle 1+: Ipatasertib + Darolutamid + ADT
  Interventions: Drug: Ipatasertib; Drug: Darolutamide; Drug: Androgen Deprivation Therapy
- Phase II: ADT + Ipatasertib + Darolutamide (Experimental): All Cycles: Ipatasertib + Darolutamide + ADT
  Interventions: Drug: Ipatasertib; Drug: Darolutamide; Drug: Androgen Deprivation Therapy

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib
Drug: Darolutamide — Darolutamide
Drug: Androgen Deprivation Therapy — ADT per institutional standards
  Other Names: ADT

SUMMARY:
This multicenter Phase I/II trial consists of two stages: a phase I stage in patients with castration resistant prostate cancer in which the recommended phase II dose will be determined for ipatasertib administered in combination with darolutamide; and a phase II neoadjuvant stage in which patients with high risk prostate cancer and loss of PI3K pathway activation in the tumor tissue planning on undergoing prostatectomy receive ADT, darolutamide, and ipatasertib for 24 weeks prior to planned surgery.

DETAILED DESCRIPTION:
The proposed trial is a single arm, two stage trial looking for an efficacy signal in the neoadjuvant setting in patients with PTEN-null tumors. The active therapy is a combination of androgen deprivation therapy, darolutamide, and ipatasertib. Patients will be treated for 6 months prior to prostatectomy, since previous studies have shown that pCR+MRD rate is higher with 6 months of ADT + abiraterone (24%) than 3 months (4%) (Taplan ME et al. J Clin Oncol. 2014;32(33):3705-15). Since the combination has not been evaluated before, a lead-in cohort in patients with castration resistant prostate cancer will be performed to evaluate safety and drug-drug interaction.

The lead-in cohort will enroll 6 patients to assess the safety of ipatasertib and darolutamide. Ipatasertib has already been evaluated in combination with the AR pathway inhibitors abiraterone and enzalutamide, where 400 mg was found to be safe. Therefore patients will receive the expected final dose of darolutamide 600 mg BID and ipatasertib 400 mg daily. Toxicities will be monitored for 28 days, and blood samples will be drawn for pharmacokinetic (PK) studies. If one or fewer patients experience a DLT the trial will advance to the neoadjuvant setting. If two or more patients experience a DLT at 400 mg, the dose will be reduced for already enrolled patients and another 6 patients will be enrolled to evaluate darolutamide 600 mg BID and ipatasertib 200 mg daily.

PK evaluations will continue for a total of 6 months. Enrollment in the neoadjuvant cohort can proceed before PK studies are complete.

Patients in the Phase I portion will have response evaluated at 12 weeks, including PSA response and radiographic response per modified PCWG3. If there is progression on bone scan alone, patients should have confirmatory bone scan at least 6 weeks later. Patients will continue on therapy until the time of progression.

ELIGIBILITY:
Eligibility Criteria Approximately 26-38 patients with prostate cancer will be enrolled in this study. This includes 6-18 patients in the Phase I de-escalation cohort with metastatic or nonmetastatic castration resistant prostate cancer, and 20 patients in the Phase II neoadjuvant cohort with high risk localized or locally advanced prostate cancer that has PI3K pathway activation.

* For the Phase I de-escalation cohort, the patient must have castration resistant prostate cancer (metastatic or non-metastatic), as defined by PCWG3.
* For the Phase II neoadjuvant cohort, the patient must be a candidate for radical prostatectomy at the time of enrollment and be planning to undergo this procedure. The patient must have a histologically-confirmed diagnosis of localized, untreated prostate cancer with high risk features and must have sufficient archival tissue (at least 2 cores) available for targeted sequencing and immunohistochemistry (IHC). The tumor must have PI3K pathway activation. This can be determined by IHC, in which case at least 50% of the tumor tissue evaluated must be negative for PTEN expression by immunohistochemistry on local review. Alternatively, qualifying alteration in PTEN, PIK3CA, or AKT1 on next generation sequencing (NGS) is also acceptable to be eligible, regardless of PTEN expression. If the patient qualifies based on NGS results, IHC must still be performed.

  * Qualifying mutations include changes in AKT1 at residues E17, L52, or Q79; in PIK3CA at residues R88, G106, K111, G118, N345, E542, E545, Q546, M1043, H1047, or G1049; in PTEN a R130Q/C/H substitution or a deletion, frameshift, or introduction of early stop codon. The assay must be a CLIA-certified assay, and a copy of the report must be provided.

Phase I Inclusion Criteria:

* Histologically confirmed prostate cancer
* Male and >= 18 years of age
* ECOG performance status of <= 2
* Castration resistant prostate cancer, defined as biochemical, radiographic, and/or clinical progression despite castrate level of testosterone (<50 ng/dL). There is no restriction on prior therapies for CRPC.
* Evaluable disease, with PSA >= 1.0 ng/ml (nmCRPC) or visible prostate cancer on imaging (mCRPC).
* Serum testosterone < 50 ng/dL
* Willing to undergo blood draws to measure PK levels
* Able to swallow pills
* Must have ability to understand and the willingness to sign a written informed consent prior to receiving a subject ID number.
* Unless surgically sterile, sexually active patients must agree to use effective barrier method and refrain from sperm donation during the study treatment and for 3 months after the end of study treatment.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 14 days prior to registration.
* Hematological

  --Hemoglobin (Hgb): >/= 9 g/dL
  * Absolute Neutrophil Count (ANC): >/= 1,500/uL
  * Platelet count: >/= 100,000/uL
* Renal --Creatinine: </= 2 x upper limit of normal (ULN)
* Hepatic

  --Bilirubin: </= 1.5 ULN or Gilbert's syndrome with normal direct bilirubin
  * Aspartate aminotransferase (AST) </= 2.5 x ULN
  * Alanine aminotransferase (ALT): </= 2.5 x ULN
* Blood sugar

  * HbA1C: </= 7.5%
  * Fasting glucose</= 150 mg/dL

Phase I Exclusion Criteria:

* Patients receiving systemic therapy for prostate cancer <= 21 days or 5 half-lives (whichever is shorter) prior to starting study drug are not eligible.

  --NOTE: Patients must continue Androgen Deprivation Therapy, and patients can receive bone supportive therapy.
* Histology of small cell carcinoma prostate cancer. Adenocarcinoma with neuroendocrine features is allowed.
* Any active infection requiring IV antibiotics
* Known additional malignancy that has a life-expectancy < 2 years.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

  * hepatitis B (known positive HBV surface antigen (HBsAg) result),
  * hepatitis C, or
  * human immunodeficiency virus (positive HIV 1/2 antibodies). ---NOTES: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for >= 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy.
* History of type I or type II diabetes mellitus requiring insulin.
* Any of the following within 6 months before registration: stroke, myocardial infarction, severe/unstable anginal pectoris, coronary/peripheral artery bypass graft, congestive heart failure New York Heart Association (NYHA) class III or IV.
* Congenital long QT syndrome or QTcF > 480 milliseconds
* Grade >= 2 uncontrolled or untreated hypercholesterolemia (>300 mg/dL) or hypertriglyceridemia (>300 mg/dL)
* History of or active inflammatory bowel disease (IBD) or active bowel inflammation (diverticulitis)
* Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug
* History of allergic reaction to darolutamide or ipatasertib.
* Any condition that in the opinion of the investigator would impair the patients' ability to comply with study procedures.

Phase II Inclusion Criteria:

-Histologically-confirmed diagnosis of localized, untreated prostate cancer with high-risk features. High-risk features is defined as:

* Two or more cores from prostate biopsy that are grade group 4 (Gleason score 4+4=8) or higher, OR
* Stage T3-4 (by clinical exam or MRI), M0, and at least 2 cores from prostate biopsy that are grade group 3 (Gleason score 4+3=7) or higher.

NOTE: Pathology confirmation of malignancy must be performed by the participating site (i.e. reports should be issued by the participating site; if a subject's pathology report was not issued by the participating site, archival tissue should be requested by the participating site for internal pathology review.)

* Sufficient archival tissue (at least 2 cores) available for targeted sequencing and immunohistochemistry to evaluate for PTEN loss using the Ventana SP218 immunohistochemistry assay at the local institution. Next generation sequencing is also acceptable to be eligible regardless of IHC result, but there must also be sufficient tissue to evaluate for PTEN by IHC.

  --The tumor evaluated for PTEN expression should be selected based on containing both high grade and high volume of tumor content. The slide evaluated for PTEN expression should be saved for confirmatory central review. Eligibility is based on local review.
* Measurable PSA
* Must have evidence of PI3K pathway activation. This can be by demonstrating PTEN loss per local institution evaluation, defined as 50% or more of tumor tissue being negative for PTEN expression on Ventana SP218 immunohistochemistry assay. Alternatively, qualifying alteration in PTEN, PIK3CA, or AKT1 on next generation sequencing is also acceptable to be eligible, regardless of PTEN expression.

  --Qualifying mutations include changes in AKT1 at residues E17, L52, or Q79; in PIK3CA at residues R88, G106, K111, G118, N345, E542, E545, Q546, M1043, H1047, or G1049; or in PTEN a R130Q/C/H substitution, or a deletion, frameshift, or introduction of early stop codon. The assay must be a CLIA-certified assay, and a copy of the report must be provided.
* Disease must be untreated and subject must be eligible for (per PI discretion) and planning to undergo radical prostatectomy.
* Male and ≥18 years of age.
* ECOG performance status of ≤ 1 within 14 days prior to signing consent.
* CT or MRI of abdomen and pelvis and bone scan within ≤90 days prior to starting study drug.
* Able to swallow pills
* Must have ability to understand and the willingness to sign a written informed consent prior to starting study drug.
* Sexually active patients, unless surgically sterile, must agree to use effective barrier method and refrain from sperm donation during the study treatment and for 3 months after the end of study treatment.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 14 days prior to registration.

Phase II Exclusion Criteria:

* Histology of small cell carcinoma prostate cancer. Adenocarcinoma with neuroendocrine features is allowed.
* Active infection requiring IV antibiotics
* Distant metastatic disease beyond N1 (regional) lymph nodes on conventional baseline imaging studies within 90 days prior to signing consent.
* Known additional malignancy that has a life-expectancy < 5 years.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

  * tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice),
  * hepatitis B (known positive HBV surface antigen (HBsAg) result),
  * hepatitis C, or
  * human immunodeficiency virus (positive HIV 1/2 antibodies). NOTES: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for ≥ 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.
* Prior treatment of prostate cancer with: second generation androgen receptor (AR) inhibitors, other investigational AR inhibitors or CYP17 enzyme inhibitor, radiation therapy, surgery, or chemotherapy. First generation antiandrogen (e.g. bicalutamide) for 28 days or fewer is allowed.
* Receipt of an investigational agent within <= 28 days prior to registration; or herbal medications and marijuana products within <= 1 day prior to registration.
* Receipt of medications (e.g. finasteride, dutasteride) or agents that are likely to alter serum PSA levels within <= 42 days or 5 half-lives prior to registration, whichever is shorter.
* History of type I or type II diabetes mellitus requiring insulin.
* Any of the following within 6 months before registration: stroke, myocardial infarction, severe/unstable anginal pectoris, coronary/peripheral artery bypass graft, congestive heart failure New York Heart Association (NYHA) class III or IV.
* Congenital long QT syndrome or QTcF > 480 milliseconds
* Grade >= 2 uncontrolled or untreated hypercholesterolemia (>300 mg/dL) or hypertriglyceridemia (>300 mg/dL)
* History of or active IBD or active bowel inflammation (diverticulitis)
* Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug
* History of allergic reaction to darolutamide or ipatasertib.
* Any condition that in the opinion of the investigator would impair the patients' ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject's must be biologically male to participate in this study
Enrollment: 6 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David VanderWeele, MD\Phd, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Penn State Cancer Institute, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT: Cycle 0 Days 1-7: Ipatasertib Monotherapy + Androgen Deprivation Therapy (ADT)
  Cycle 1 Day 1+: Ipatasertib 400 mg daily (AM dose with PKs)+ Darolutamide 600 mg BID (No AM dose.PM dose taken after ipatasertib monotherapy PKs)+ ADT (per institutional standards)
- Phase I De-Escalation Cohort, Level -2: Ipatasertib 200 mg Daily + Darolutamide 600 mg BID + ADT: Cycle 0 Days 1-7: Ipatasertib Monotherapy + Androgen Deprivation Therapy (ADT)
  Cycle 1 Day 1+: Ipatasertib 200 mg daily (AM dose with PKs)+ Darolutamide 600 mg BID (No AM dose.PM dose taken after ipatasertib monotherapy PKs)+ ADT (per institutional standards)
- Phase I De-Escalation Cohort, Level -2: Ipatasertib 300 mg Daily + Darolutamide 600 mg BID + ADT: Cycle 0 Days 1-7: Ipatasertib Monotherapy + Androgen Deprivation Therapy (ADT)
  Cycle 1 Day 1+: Ipatasertib 300 mg daily (AM dose with PKs)+ Darolutamide 600 mg BID (No AM dose.PM dose taken after ipatasertib monotherapy PKs)+ ADT (per institutional standards)
- Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT: All Cycles: Ipatasertib + Darolutamide + ADT
  Ipatasertib: Ipatasertib were planned to be administered orally per Phase I cohort determined dose of 400mg daily for each cycle length of 28 days
  Darolutamide: Darolutamide were planned to be administered orally at a dose of 600mg BID for each cycle length of 28 days
  Androgen Deprivation Therapy: ADT per institutional standards
Period: Study Treatment
Arm/Group | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT | Phase I De-Escalation Cohort, Level -2: Ipatasertib 200 mg Daily + Darolutamide 600 mg BID + ADT | Phase I De-Escalation Cohort, Level -2: Ipatasertib 300 mg Daily + Darolutamide 600 mg BID + ADT | Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT
Started | 6 | 0 (No subjects were enrolled at this level.) | 0 (No subjects were enrolled at this level.) | 0 (Study was terminated before subjects were enrolled at Phase II due to Funder's Decision.)
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Disease Progression | 5 | 0 | 0 | 0
Not completed — Death on study | 1 | 0 | 0 | 0
Period: Follow up
Arm/Group | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT | Phase I De-Escalation Cohort, Level -2: Ipatasertib 200 mg Daily + Darolutamide 600 mg BID + ADT | Phase I De-Escalation Cohort, Level -2: Ipatasertib 300 mg Daily + Darolutamide 600 mg BID + ADT | Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 5 (One subject died on treatment.) | 0 (No subjects were enrolled at this level.) | 0 (No subjects were enrolled at this level.) | 0 (Study was terminated before subjects were enrolled at Phase II due to Funder's Decision.)
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [60.8 to 70.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Gleason score [Count of Participants; unit: Participants] — A 5 Grade Group System was created to have a better way to describe how a cancer will behave and respond to treatment.
  Grade group 1: Gleason score 6 or lower (low-grade cancer) Grade group 2: Gleason score 3 + 4 = 7 (medium-grade cancer) Grade group 3: Gleason score 4 + 3 = 7 (medium-grade cancer) Grade group 4: Gleason score 8 (high-grade cancer) Grade group 5: Gleason score 9 to 10 (high-grade cancer)
  Participants
    Gleason Score 3 | 2
    Gleason score 4 | 1
    Gleason score 7 | 3
Tumor Location [Count of Participants; unit: Participants]
  Acinar Adenocarcinoma | 1
  Adenocarcinoma NOS | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Pathological Complete Response (pCR) Rate
Description: Combined rate of pathologic complete response (pCR) (defined as absence of pathologic disease on hematoxylin and eosin (H&E) stain (ypT0)), or with presence of minimal residual disease (<5 mm linearly)
Time Frame: From C1D1 until death.
Population: Study was terminated after the completion of Phase I accrual. No data for this cancelled Phase II objective was collected or analyzed as no prostatectomies were performed in any subject (a pre-requisite for determining pCR).
Arm/Group | Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT
Number analyzed (Participants) | 0

2. Secondary Outcome: Summary of Dose-Limiting Toxicities
Description: A summary of all dose-limiting toxicities experienced by Phase I subjects within the first cycle (28 days) of treatment, as defined in the study protocol.
Time Frame: Until the completion of cycle 1, 28 days
Population: Six Phase I subjects are included in the analysis population.
Measure: Number; unit: dose-limiting toxicities
Groups:
- Phase I De-Escalation Cohort: All Cycles: Ipatasertib 400mg + Darolutamide 600mg BID + ADT per institutional guidelines
Arm/Group | Phase I De-Escalation Cohort
Number analyzed (Participants) | 6
dose-limiting toxicities | 0

3. Secondary Outcome: Phase II - Two Year Biochemical Recurrence-free Survival
Description: Two year biochemical recurrence-free survival (PSA ≤ 0.2 ng/mL) will be measured in men with high risk, localized, prostate cancer that is lacking PTEN
Time Frame: From C1D1 until death or up to a maximum of 24 months
Population: Study was terminated after the completion of Phase I accrual. No Phase II subjects were accrued, and no data for this cancelled Phase II objective were collected or analyzed. Additionally, no subjects from the Phase I study were followed for sufficient time to collect two-year biochemical recurrence-free survival, as they did not consent for this activity.
Arm/Group | Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase II: Rate of PSA0
Description: Rate of PSA0 (undetectable PSA on local institutions laboratory testing with testosterone recovery and no additional therapy) will be measured in men with high risk, localized, prostate cancer that is lacking PTEN.
Time Frame: From C1D1 until death.
Population: Study was terminated after the completion of Phase I accrual. No Phase II subjects were accrued, treated, or evaluated for this objective, and no data for this cancelled Phase II objective was collected or analyzed. This analysis was planned in only Phase II subjects.
Arm/Group | Phase II Neoadjuvant Cohort,MTD: Ipatasertib 400 mg + Darolutamide 600 mg BID + ADT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of consent for at least 30 days after treatment discontinuation or until a new anti-cancer treatment starts, whichever occurs first or up to a maximum of 8 months.
Description: Adverse events were recorded from the time of consent for at least 30 days after treatment discontinuation or until a new anti-cancer treatment starts, whichever occurs first, per Common Terminology Criteria for Adverse Events (CTCAE) v5.
Arm/Group | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT (N=6)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I De-Escalation Cohort, Level 1: Ipatasertib 400 mg Daily + Darolutamide 600 mg BID + ADT (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (7)
ANEMIA (Blood and lymphatic system disorders) | 6 (12)
ANOREXIA (Metabolism and nutrition disorders) | 4 (9)
ANXIETY (Psychiatric disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2)
ATAXIA (Nervous system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 5 (24)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1)
CHILLS (General disorders) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (4)
CREATININE INCREASED (Investigations) | 2 (3)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 5 (12)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
EYE DISORDERS (Eye disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 5 (8)
FEVER (General disorders) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (12)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 3 (4)
INVESTIGATIONS (Investigations) | 5 (20)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (9)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 3 (11)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (6)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERIPHERAL NERVE INFECTION (Infections and infestations) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 2 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (2)
RECURRENT LARYNGEAL NERVE PALSY (Nervous system disorders) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 3 (3)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04737109/Prot_SAP_000.pdf